CLINICAL TRIAL: NCT01524692
Title: A Phase II Pilot Study of Dovitinib (TKI258) in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma.
Brief Title: Study of Dovitinib (TKI258) in Adenoid Cystic Carcinoma
Acronym: ACC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Patrick Dillon, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15627
Record Dates: First submitted 2012-01-17; First posted 2012-02-02 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single ARM Dovitinib treatment (Experimental): Single ARM Dovitinib treatment
  Interventions: Drug: Dovitinib (TKI258)

INTERVENTIONS:
Drug: Dovitinib (TKI258) — 500 mg orally on a 5-days on/2-days off schedule each week of a 4-week (28-day) cycle. Treatment will continue until progression as defined by RECIST, unacceptable adverse events, patient refusal to continue on study, or physician's decision to withdraw the patient.

SUMMARY:
The purpose of this study is to improve survival of patients with recurrent or metastatic Adenoid Cystic Carcinoma (ACC). This study will test the efficacy of the investigational drug, TKI258, in treating ACC.

DETAILED DESCRIPTION:
Adenoid cystic carcinoma (ACC) is an uncommon malignancy that arises in secretory glands. The most common sites for the disease are the major and minor salivary glands but these tumors may also arise in the nasal cavity, lacrimal gland, tracheobronchial tree, breast or vulva. The mainstay of treatment for localized ACC is surgical resection often followed by post-operative radiotherapy. Although this leads to an initially high rate of local control, the 5-year disease-free survival rate is 50-75%. In addition, a significant proportion of the patients develop distant metastases, most frequently in the lung. Compared to other malignancies, ACC tends to grow more slowly. Thus, patients often do well in the short-term but long-term prognosis remains guarded and most succumb to the disease within 10-15 years. To date, systemic therapies have proven to be largely ineffective against recurrent and metastatic ACC. Dovitinib is a broad-targeted-profiled RTK inhibitor active against these three RTKs (VEGF, FGF and PDGF) involved in tumor cell growth. Based on its potency as an inhibitor of these RTKs both in vitro and in vivo, and the compound's oral availability, several clinical trials of dovitinib are underway. This phase II trial will test the hypothesis that dovitinib will be active against this disease. The rationale is based on pre-clinical studies that suggest that dovitinib suppresses tumor growth by blocking constitutive signaling of the fibroblast growth factor receptor-1 (FGFR1) and animal studies in which the drug proved to be active against primary ACC xenografts.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. Patients must have histology or cytology studies that confirm the diagnosis of adenoid cystic carcinoma. (Note: Subsequent central review of the pathology slides will be provided by Drs. Christopher Moskaluk or Henry Frierson, Department of Pathology at the University of Virginia Health Sciences Center).
2. Patients must have recurrent and/or metastatic disease that is not amenable to potentially curative surgical resection or radiotherapy.
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with spiral CT scan (or >20 mm with conventional techniques). Pathologic lymph nodes are measured by shortest diameter as per RECIST.
4. Patients must have serial imaging that allows measurement of tumor growth rates by change point analysis:

1. The remote baseline study scan must be within six calendar months of the immediate pre-study scan.

2. The remote baseline scan must have measurable disease ≥ 10 mm for non-pulmonary lesions or ≥ 4 mm for pulmonary metastases that show subsequent progression.

3. Comparison of the remote baseline and subsequent studies must show progressive disease in 1-5 selected target lesions based on the following:

1. Modified RECIST criteria (i.e. proportional increase of 1.2 or the appearance of new lesions) AND/OR
2. Progression by change point analysis with an increase in the slope of the average tumor measurements of at least 0.22 b

a = "remote baseline scan" refers to scan done prior to pre-study scan which is used to determine pre-treatment tumor growth rate.

b = the estimated mean minus one standard deviation based on analysis of progressive tumors from untreated patients with ACC.

5. Life expectancy > 16 weeks.

6. ECOG (WHO) performance status 0-2

7. Age ≥ 18 years old

8. Patients must have the following laboratory values:

* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin (Hgb) > 9 g/dL
* Serum total bilirubin: ≤ 1.5 x ULN
* ALT and AST ≤ 3.0 x ULN
* Serum creatinine ≤ 1.5 x ULN or serum creatinine >1.5 - 3 x ULN if calculated creatinine clearance (CrCl) is ≥ 30 mL/min using the Cockroft-Gault equation, see formula below:

CrCl = [140-age (years)] x weight (kg) / [72 x serum Cr (mg/dL)] (if patient is female multiply the above by 0.85)

9. Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

Patients are ineligible for this study if he or she has any of the following:

1. Patients with brain metastases
2. Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer)
3. Patients who have received the last administration of an anticancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosurea, mitomycin-C, targeted therapy and radiation) ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
4. Patients who have received the last administration of nitrosurea or mitomycin-C ≤ 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
5. Patients who have received targeted therapy (e.g. sunitinib, sorafenib, pazopanib) ≤ 2 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
6. Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug or ≤ 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture), if the measurable lesions are outside the radiation field. Also excluded would be those who have not recovered from toxicity radiotherapy.
7. Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
8. Patients with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

   * Impaired cardiac function or clinically significant cardiac diseases, including any of the following:
   * History or presence of serious uncontrolled ventricular arrhythmias
   * Clinically significant resting bradycardia
   * LVEF assessed by 2-D echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) < 45%
   * Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)
   * Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s)

     1. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
     2. Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
     3. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
     4. Patients who are currently receiving anticoagulation treatment with therapeutic doses of warfarin
     5. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
9. Pregnant or breast-feeding women
10. Women of child-bearing potential not employing an effective method of birth control. Two birth control methods must be used throughout the trial and one month after the last dose of study drug (e.g. condom with spermicidal jelly, foam suppository or film; diaphragm with spermicide; male condom and diaphragm with spermicide). Contraceptives that are affected by cytochrome P450 interactions (e.g. oral, implantable, injectable, or intrauterine hormonal contraceptives) are not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 7 days prior to starting study drug.
11. Fertile males not willing to use contraception, as stated above
12. Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single ARM Dovitinib Treatment
Started | 35
Completed | 32
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single ARM Dovitinib Treatment
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 1
  Unknown or Not Reported | 1
ECOG Performance Status [Mean (Full Range); unit: units on a scale] — ECOG PERFORMANCE STATUS
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  units on a scale | 1 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Determine the Objective Tumor Response Rate Following Treatment With TKI258
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by cross sectional imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From enrollment up to 36months
Population: 1 patient was not evaluable for response evaluation due to withdrawal prior to first interval scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Single ARM Dovitinib Treatment
Number analyzed (Participants) | 34
Participants
  Partial Response | 2
  Stable Disease | 22
  Progressive Disease | 10

2. Secondary Outcome: Estimate the Progression-free Survival Following Treatment With TKI258.
Description: PFS is measured from enrollment up to first progression event (median= 8.2 months). 1 patient was not evaluable for response evaluation due to withdrawal prior to first interval scan.
Time Frame: From enrollment up to first progression event
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Single ARM Dovitinib Treatment
Number analyzed (Participants) | 34
Months | 8.2 [7.3 to 11.0]

3. Secondary Outcome: The Adverse Event Profile of TKI258 in Subjects Who Have ACC.
Description: Adverse events were collected per CTCAE v3.
Time Frame: From enrollment up to 36months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Any Adverse Event: Patients with any adverse event as defined by CTCAE
Arm/Group | Patients With Any Adverse Event
Number analyzed (Participants) | 35
Participants | 35

4. Secondary Outcome: Quality of Life Measurements During TKI258 Treatment.
Description: Participants were asked to fill out FACT-G (Functional Assessment of Chronic Illness Therapy) quality of life questionnaires at baseline and off-treatment visit (average 8.2 months). This scale measures physical well-being, social/family well-being, emotional well-being, and functional well-being on a 5 point Likert scale. Scores range from 0 to 4 on a Likert scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The raw score range for each subscale is 0-28 points and the total score range is 0-108. Higher values represent higher well-being in each functional subscale. The mean difference from baseline to off-study assessment are presented with range from minimum to maximum.
Time Frame: Baseline FACT-G questionnaire and FACT-G questionnaire at time of off-treatment visit (average of 8.2 months)
Population: All participants filled out quality of life questionnaires.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Single ARM Dovitinib Treatment
Number analyzed (Participants) | 35
units on a scale
  Functional Well-being subscale mean difference | -4 [-12 to -1]
  Physical Well-being subscale mean difference | -6 [-18 to 7]
  Social Well-being mean Difference | -1 [-10 to 28]
  Emotional Well-being mean Difference | -3 [-12 to 11]
  Overall FACT-G mean difference | -13 [-44 to 20]

5. Secondary Outcome: Feasibility of Measuring and Analyzing TKI258 Induced Changes in the Growth Rate of Adenoid Cystic Carcinomas.
Description: Collect descriptive data about the change in tumor growth rates as measured by the change point method. Tumor growth rate is defined as the estimated slope (slope is then defined as Y1-Y0 divided by X1-X0) from tumor measurements taken prior to treatment (TG0). TG0 is compared with TG1 (tumor growth rate) as defined by the estimated slope after treatment (comparing time 0 to 4mo). Each patient's tumor growth profile is allowed one slope measured from pre-study (-6 months to time 0), and the other slope (time 0 to time 4 months). Change between those 2 slopes is reported. Slope is measured on a plot of time on the x axis and sum of longest diameters of RECIST target lesions on the y axis. The slope of the tumor growth curve (plotted as sum of longest diameters vs month since starting dovitinib) is measured at time points -6mo, 0, and 4 months. Pre-study scans (-6mo) were required of all patients and on-study scans were at times, 0, 2, 4months, 8months, 12mo, 16mo.
Time Frame: All patients provided pre-study scans with target lesions. The target lesions from pre-study scans were compared to the target lesions on the baseline scan at time 0. TG0 was measured from -6 months to time 0. TG1 is defined as time 0 to time 4 months.
Population: All treated patients were required to submit pre-study cross sectional imaging from preceeding 6months in order to establish pre-study tumor growth rates. On-study scans were performed at time 0, 2, 4 months, 8, months, 12 months, 16 months.
Measure: Mean (Standard Error); unit: cm/month
Arm/Group | Single ARM Dovitinib Treatment
Number analyzed (Participants) | 35
cm/month
  Slope of Tumor growth rate from -6mo to time 0 | 1.95 (0.29)
  Slope of tumor growth rate from 0 to 4 months | 0.63 (0.18)

6. Secondary Outcome: Expression of MYB Protein and Chromosomal Rearrangements of the MYB Locus
Description: Assess archival tumor samples for the expression of MYB protein and chromosomal rearrangements of the MYB locus.
Time Frame: Anticipated Reporting Date 2020
Reporting Status: Not Posted, anticipated posting 2020-12

ADVERSE EVENTS:
Time Frame: AE's and SAE's were collected from date of consent until off study date (which ranged from 0-20 months). Overall survival was collected from time of consent to June 2015 (40 months.)
Description: AE reporting was completed using CTCAE 4.03
Arm/Group | Single ARM Dovitinib Treatment
All-Cause Mortality (participants affected / at risk) | 16/35
Serious Adverse Events (participants affected / at risk) | 22/35
Other Adverse Events (participants affected / at risk) | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single ARM Dovitinib Treatment (N=35)
Anemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 1
Stomach Pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
GGT Elevation (Hepatobiliary disorders) | 4
Dehydration (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hypertriglyceridemia (Hepatobiliary disorders) | 9
Anxiety (Psychiatric disorders) | 1
Thromboembolic Event (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Pain (General disorders) | 2
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single ARM Dovitinib Treatment (N=35)
Anemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 1
Stomach Pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
GGT Elevation (Hepatobiliary disorders) | 4
Dehydration (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 1
Thromboembolic Event (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Pain (General disorders) | 2
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No